CLINICAL TRIAL: NCT04645810
Title: A Pilot Study of Focal Salvage High-Dose-Rate Brachytherapy for Prostate Gland Only Recurrence
Brief Title: A Study of Focal Salvage High-Dose-Rate Brachytherapy for Prostate Gland Only Recurrence
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study stopped early, did not enroll anyone, and will not resume
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Hong Zhang, Associate Professor - Department of Radiation Oncology (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005667
Record Dates: First submitted 2020-11-22; First posted 2020-11-27 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer; HDR
Keywords: Brachytherapy; Prostate Cancer; High-Dose-Rate (HDR)
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: High-Dose-Rate prostate brachytherapy (Experimental): High-Dose-Rate brachytherapy, 2 fractions
  Interventions: Procedure: High-Dose-Rate Brachytherapy

INTERVENTIONS:
Procedure: High-Dose-Rate Brachytherapy — High-Dose-Rate Brachytherapy Targeting only to AXUMIN PET Visible Lesion

SUMMARY:
The purpose of this study is to learn more about what effects the use of high-dose-rate (HDR) brachytherapy on prostate cancer recurrence, seen by AXUMIN PET scan, has on prostate cancer.

DETAILED DESCRIPTION:
In this study the investigator would like to better understand the use of high-dose rate (HDR) brachytherapy to target only recurrent prostate cancer that can be seen by AXUMIN PET scan. The use of HDR brachytherapy for prostate cancer is not new, but it is a more recent advancement to use it to treat only what can be seen instead of the whole prostate.

ELIGIBILITY:
Inclusion Criteria:

History of histologically confirmed, clinically localized adenocarcinoma of the prostate treated with external beam radiation, brachytherapy, or combination of external beam radiation and brachytherapy, with curative intent completed at least 24 months ago F-18 fluciclovine (AXUMIN) PET scan within 90 days prior to registration demonstrating recurrent lesion within the prostate gland Biopsy confirmation of disease recurrence within the prostate gland Age ≥ 18 KPS ≥ 70% Suitable candidate for brachytherapy based on established criteria IPSS score <16 No pelvic arch interference No Rectal fistula/fissure Fit for general or spinal anesthesia No history of urethral stricture Ability to understand, and willingness to sign the written informed consent

Exclusion Criteria:

Evidence of metastatic or nodal disease outside of the prostate gland on AXUMIN PET scan within 90 days prior to enrollment Patient unable to have MRI Patients with neuroendocrine or small cell carcinoma of the prostate TURP within 6 months prior to enrollment History of Crohn's disease, ulcerative colitis, or known radiation proctitis Inability to understand spoken and written English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with prostate-specific antigen (PSA) levels rising of 2ng/ml or above | 6 Months
  Rate of prostate-specific antigen (PSA) failure after focal salvage HDR in the setting of prostate only recurrence after primary non-surgical treatment, defined as a PSA rise of 2 ng/ml or more above the nadir at 6 months
Incidence of Treatment-Related Adverse Events [Safety and Tolerability] | 6 Months
  Measured by adverse event severity and quantity

SECONDARY OUTCOMES:
Progression Free Survival | 6 Months
  Measure of time from study enrollment until progression.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, Principal Investigator — University of Rochester Wilmot Cancer Center
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No